CLINICAL TRIAL: NCT05501600
Title: Neural Correlates of Lidocaine Analgesia
Acronym: NeuCLA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keith M Vogt (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor-Investigator, Keith M Vogt, Associate Professor of Anesthesiology & Perioperative Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21120115; R35GM146822 (NIH)
Record Dates: First submitted 2022-08-02; First posted 2022-08-15 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia; Pain
Keywords: lidocaine; functional MRI; electric nerve stimulation; functional connectivity
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lidocaine (Experimental): Subjects will receive lidocaine during the drug portion of the experiment.
  Interventions: Device: Peripheral Nerve Stimulation; Drug: Lidocaine IV

INTERVENTIONS:
Device: Peripheral Nerve Stimulation — Experimental acute pain stimulus will be delivered using an electric nerve stimulator.
  Other Names: Electric Nerve Stimulation
Drug: Lidocaine IV — Subjects will receive an intravenous infusion of lidocaine for about 30 minutes.
  Other Names: Xylocaine

SUMMARY:
The purpose of this study is to characterize the effects of intravenous lidocaine on pain processing and cognitive function. Functional magnetic resonance imaging will be used to identify the neural correlates of these phenomena. The study will consist of 1 visit and involves no long-term follow up.

DETAILED DESCRIPTION:
This is an observational cohort study of volunteer subjects, which will employ neuroimaging and behavioral measures to characterize the effects of intravenous lidocaine on pain processing and cognitive function. A steady-state effect-site concentration of lidocaine will be achieved, and a short battery of cognitive behavioral tasks will be employed. At the dose target, pain task functional MRI and resting-state connectivity will be determined. This work will use a systems neuroscience approach to fill an important knowledge gap about the central effects of intravenous lidocaine, a commonly-used opioid alternative analgesic agent.

Aim1: Determine cognitive behavioral effects of a steady-state dose of IV lidocaine using a short battery of tasks. The investigators hypothesize that the administration of lidocaine will correlate to decreased pain ratings, slowed psychomotor response, and decreased memory encoding.

Aim2: Determine the neural effects of a steady-state dose of IV lidocaine in response to acute pain, and on resting connectivity. The investigators hypothesize that pain task-related activation will decrease in the insula and anterior cingulate, corresponding to decreased ratings of pain intensity and unpleasantness. Additionally, the investigators expect widespread decreases in long-range functional connectivity between brain areas know to be involved in these two areas and other known to be involved in pain processing.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70
* Be of normal body-weight
* Be generally healthy
* Have none of the specific exclusion criteria
* Have a valid email address and phone number throughout the study

Exclusion Criteria:

* Pregnancy
* Body mass index > 40
* Having moderate to severe sleep apnea
* Having chronic pain requiring the regular use of pain medicine 3 or more times per week
* Having neurologic or psychiatric disease, including benign tremor, anxiety, and depression
* Having a history of seizures
* Having history of cardiac rhythm disturbance (such as heart block, or atrial fibrillation)
* Being severely claustrophobic
* Having metal implants or non-removable metal piercings
* Having metal-containing tattoos, particularly on the face
* Having a history of adverse reaction to lidocaine
* Are regularly taking: antiepileptics, antidepressants, anti-psychotics, anti-anxiety medication, stimulants, sleep-aids, or pain medication
* Are taking prescribed medications for psychiatric or neurological conditions
* Having hypersensitivity to lidocaine or to any other local anesthetics of the amide type
* Having Wolff-Parkinson-White syndrome
* Having known renal or hepatic dysfunction
* having glucose-6-phosphate dehydrogenase deficiency or history of methemoglobinemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Vogt, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vogt KM, Burlew AC, Simmons MA, Reddy SN, Kozdron CN, Ibinson JW. Neural correlates of systemic lidocaine administration in healthy adults measured by functional MRI: a single arm open label study. Br J Anaesth. 2025 Feb;134(2):414-424. doi: 10.1016/j.bja.2024.07.039. Epub 2024 Oct 21. PMID 39438214

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine
Started | 30
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Completed participants
Groups:
- Lidocaine: Subjects receiving lidocaine during the drug portion of the experiment.
Arm/Group | Lidocaine
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 1
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Brain Activation to Painful Stimulation Difference: Drug-free Condition Minus Lidocaine Condition
Description: The Z-score is calculated by linear regression of the task timing against the MRI signal time-course (MRI data is in arbitrary units with no maximum or minimum) at each voxel (single data point in brain). Primary outcome is listed for the Right insula, but similar scores are calculated throughout the brain. Z-score of 0 indicates no task-related changes. Z-scores further from zero indicate stronger correlation between functional MRI signal change and the task timing, with positive values indicating increases in fMRI signal and negative Z-scores indicating decreases. Practically, higher positive Z-scores indicate increased brain activity and larger negative Z-scores indicate decreased brain activity. This outcome is reported as a number, as it is calculated using all the data across subjects combined into one statistical measure for the overall strength of difference in MRI signal change between two groups of data. Dispersion measures cannot be calculated for the summary Z-score.
Time Frame: 4.5 minutes
Measure: Number; unit: Z-score
Arm/Group | Lidocaine
Number analyzed (Participants) | 27
Z-score | 3.6
Statistical Analysis 1: Comparison: Lidocaine; Test type: Superiority; p = 0.004, Regression, Linear

2. Primary Outcome: Resting-state Functional Connectivity Difference: Drug-free Minus Lidocaine
Description: Functional connectivity (FC) measures the correlation of MRI signal time-series between brain regions. Changes in FC reflect differences in brain state, in this case between drug-free and lidocaine conditions. The reported value is the FC change between the right insula and anterior cingulate. A T-statistic of 0 indicates no change; more positive scores mean stronger connectivity in the drug-free condition, and more negative scores mean stronger connectivity with lidocaine. This outcome is a number reflecting the overall magnitude of difference between two datasets, calculated in one summary statistic. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.
Time Frame: 8 minutes
Measure: Number; unit: T-statistic
Arm/Group | Lidocaine
Number analyzed (Participants) | 27
T-statistic | 3.25
Statistical Analysis 1: Comparison: Lidocaine; Test type: Superiority; p = 0.081616, t-test, 2 sided

3. Secondary Outcome: Pain Intensity Score Difference, Drug-free Condition Minus Lidocaine Condition
Description: Numerical rating scale (0-10) pain score difference, comparing drug-free to the steady-state dose of lidocaine. Higher pain scores indicate more pain; a positive difference between pain score during the drug-free condition minus the value during the lidocaine condition indicates pain reduction (a better outcome).
Time Frame: 12 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine
Number analyzed (Participants) | 27
units on a scale | 0.4 (0.2)

4. Secondary Outcome: Memory Performance Difference, Drug-free Minus Lidocaine Condition
Description: Performance on a short computer-based test of memory for visual pictures will be quantified using signal detection metric d-prime, reflecting ability (in standard deviation units) to detect previously-seen images from the background "noise" of previously un-seen images. Differences will be determined between the drug-free condition and the lidocaine condition. Higher values of d-prime indicate stronger memory performance; a positive difference for drug-free minus lidocaine condition would indicate the expected decrease in memory performance.
Time Frame: 3 minutes
Measure: Mean (95% Confidence Interval); unit: d-prime
Arm/Group | Lidocaine
Number analyzed (Participants) | 27
d-prime | 0.48 [0.12 to 0.85]

5. Secondary Outcome: Motor Response Time Differences
Description: Response times (in ms) after hearing a tone will be recorded and compared between the drug-free and Lidocaine condition, with the calculated difference in response times reported. Higher values will reflect slower responses, which are expected under the lidocaine condition.
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Lidocaine
Number analyzed (Participants) | 27
milliseconds | 10 (100)

ADVERSE EVENTS:
Time Frame: 1 hour
Description: Adverse events during the experiment
Arm/Group | Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT05501600/Prot_001.pdf
  • Informed Consent Form (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT05501600/ICF_000.pdf